CLINICAL TRIAL: NCT01078701
Title: Randomised, Double-blind, Placebo-controlled, Phase IIa Dose Finding Study of Single Dose GHB11L1 in Healthy Adults
Brief Title: Dose Finding Study of Single Dose GHB11L1 in Healthy Adults
Acronym: GHB-CS07
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AVIR Green Hills Biotechnology AG (Industry)
Responsible Party: Thomas Muster PhD, CEO/CSO, AVIR Green Hills Biotechnology AG
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GHB-CS07; EudraCT 2009-015902-20 (Other: EMEA)
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2011-01

CONDITIONS: Influenza, Human
Keywords: live attenuated flu vaccines; Influenza A (H1N1); intranasal application; replication-deficient influenza virus
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GHB11L1 (Experimental): Dose levels: 6.0 log10 TCID50/volunteer, 6.5 log10 TCID50/volunteer and 7.0 log10 TCID50/volunteer
  Interventions: Biological: GHB11L1
- SPGN buffer (Placebo Comparator): SPGN buffer administration by liquid nasal spray
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: GHB11L1 — GHB11L1 administration by liquid nasal spray at doses of 6.0 log10, 6.5 log10 and 7.0 log10 TCID50/volunteer
  Other Names: A/Brisbane/59/07(H1N1)-like delNS1 virus reassortant
  Arms: GHB11L1
Biological: Placebo — SPGN buffer
  Other Names: SPGN buffer
  Arms: SPGN buffer

SUMMARY:
The purpose of this phase IIa trial is to evaluate the immunogenicity of a single dose of GHB11L1 administered by liquid nasal spray for vaccination against influenza A (H1N1) virus.

This study is also performed to assess safety, tolerability and pharmacokinetics (shedding) of a single dose of GHB11L1 administered by liquid nasal spray.

DETAILED DESCRIPTION:
GHB11L1 intends to provide a novel vaccination for influenza virus infection. 48 healthy volunteers will be included in this phase IIa study investigating three dose levels. 16 subjects will be randomised at a ratio of 3:1 for GHB11L1 or placebo.

Healthy male volunteers, 18-50 years of age and seronegative with respect to the applied virus antigens (antibody titers <1:10 detected) will be randomised.

GHB11L1 will be administered once on day 1. Follow-up visits will be performed on days 2, 8 and 29.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, 18-50 years
* Seronegative for H1N1 (Influenza A/Brisbane/59/07 antibody titres <1:10 detected in haemagglutination inhibition assay)
* Written informed consent to participate in this study

Exclusion Criteria:

* Acute febrile illness (>37.0°C)
* Signs of acute or chronic upper or lower tract respiratory illnesses (sneezing, cough, tonsillitis, otitis etc.)
* History of severe atopy
* Seasonal influenza vaccination in 2007/2008 and/or later seasons and/or pandemic influenza vaccination at any time
* Known increased tendency of nose bleeding
* Volunteers with clinically relevant abnormal paranasal anatomy
* Volunteers with clinically relevant abnormal laboratory values
* Simultaneous treatment with immunosuppressive drugs incl. Corticosteroids (≥2 weeks) within 4 weeks prior to study medication application
* Clinically relevant history of renal, hepatic, GI, cardiovascular, haematological, skin, endocrine, neurological or immunological diseases
* History of leukaemia or cancer
* HIV or Hepatitis B or C seropositivity
* Volunteers who underwent rhino or sinus surgery, or surgery of another traumatic injury of the nose within 30 days prior to application of study medication
* Volunteers who have received antiviral drugs, treatment with immunoglobulins or blood transfusions, or an investigational drug within four weeks prior to study medication application
* Volunteers who have received anti-inflammatory drugs 2 days prior to study medication application
* Volunteers who are not likely to cope with the requirements of the study or with a significant physical or mental condition that may interfere with the completion of the study

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2009-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Local and systemic immune response | From baseline to day 29 (end of study)

SECONDARY OUTCOMES:
Clinical signs and symptoms, laboratory tests Pharmacokinetics: qualitative assessment of viral recovery (shedding) in nasal mucosal samples. | From written informed consent to 30 days after end of study

CONTACTS AND LOCATIONS:
Overall Officials: Volker Wacheck, MD, Principal Investigator — Medical University Vienna
Locations (1):
- Medical University Vienna, Department of Clinical Pharmacology, Vienna, Austria